CLINICAL TRIAL: NCT01116375
Title: Does Treating Obstructive Sleep Apnea in Obese Canadian Youth Improve Blood Sugar Control? A Multi-Centered Prospective Cohort Study
Brief Title: Does Treating Obstructive Sleep Apnea in Obese Canadian Youth Improve Blood Sugar Control?
Acronym: IMPACT Obesity
Status: Completed | Type: Observational
Sponsor: Katz, Sherri Lynne, M.D. (Individual)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Dr. Sherry Lynn Katz, Katz, Sherri Lynne, M.D., Children's Hospital of Eastern Ontario
Other Study IDs: 1234
Record Dates: First submitted 2010-04-30; First posted 2010-05-05 (Estimated); Last update posted 2018-03-09 (Actual); Status verified 2018-03

CONDITIONS: Obesity; Obstructive Sleep Apnea
Keywords: Obesity; OSA; PAP therapy
MeSH Terms: conditions — Obesity; Sleep Apnea, Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Obese children with OSA: To determine whether, in obese children with moderate-severe OSA who are prescribed PAP therapy, increased hours of PAP usage per night over a one-year period is associated with a greater improvement in HOMA-IR

SUMMARY:
To determine whether, in obese children with moderate-severe Obstructive Sleep Apnea who are prescribed Positive Airway Pressure(PAP) therapy, increased hours of PAP usage per night over a one-year period is associated with a greater improvement in HOMA-IR

DETAILED DESCRIPTION:
Rationale: The five-fold increase in prevalence of childhood obesity in Canada over the last 15 years has led to an increasing number of pediatric cases of obesity-related obstructive sleep apnea (OSA). Not only is the prevalence of OSA significantly higher among obese children compared with the general population, but in this group, routine treatment by adenotonsillectomy has a much lower cure rate. Instead, Positive Airway Pressure (PAP) treatment is usually prescribed. Other complications of obesity are also increasingly recognized in children, including metabolic disturbances with insulin resistance (IR). This is particularly concerning, since IR is an identified surrogate measure of future obesity-related sequelae, such as diabetes, dyslipidemia, cardiovascular disease (including hypertension, and heart rate disturbances), inflammation and impaired quality of life. Of particular interest, the IR related to obesity can be exacerbated by OSA and the severity of IR correlates with the severity of OSA. IR is measured using a homeostasis model assessment of insulin resistance (HOMA-IR) and is calculated from fasting blood glucose and insulin levels. In obese adults with OSA, HOMA-IR, as well as cardiovascular and other metabolic markers, has been shown to improve following PAP therapy. Such a study has not been done in children. We hypothesize that PAP treatment for obese children with moderate-severe OSA will improve markers of obesity-related disease.

Primary Objective: To determine whether, in obese children with moderate-severe OSA who are prescribed PAP therapy, increased hours of PAP usage per night over a one-year period is associated with a greater improvement in HOMA-IR. Secondary Objectives: To determine whether increased hours of PAP usage per night is associated with a greater improvement in the following outcomes: 1) sympathetic nervous system activation (systolic and diastolic hypertension, nocturnal hypertension, heart rate and heart rate variability); 2) inflammation 3) neurobehavioral and quality of life measures. Methods: Study design: prospective multi-centre cohort study. Study Population: Obese children (body mass index (BMI) ≥ 95th %ile for age and sex) 8-17 years old with moderate-severe OSA will be recruited for this study from four pediatric tertiary care centres across Canada. As per current standard of care, those children with moderate-severe OSA, defined as ≥ 10 obstructive events per hour on polysomnography, will be prescribed PAP treatment. Sample Size: We expect a medium effect size (0.5); therefore 10 subjects per parameter tested (n=4) in the regression model and 25% attrition requires the recruitment of 54 subjects. Measurements will be made at baseline and 12 months. Data collection will include HOMA-IR, 24-hr blood pressure measurements, electrocardiogram for heart rate and heart rate variability, C-reactive protein as a marker of inflammation, neurobehavioral/quality of life measures (Conners parent and teacher scales, Child Behavior Checklist and Pediatric Quality of Life Inventory) and physical activity questionnaire (Habitual Activity Estimation Scale (HAES)). Data Analysis: Multivariate linear regression analyses will be performed for our primary and secondary outcomes. Our dependent variable will be change in HOMA-IR; our primary independent variable will be average number of hours/night of PAP usage. Adjustment variables will be change in BMI %ile, pubertal stage (Tanner stage 1-2 vs.

3-5), and change in HAES. Similar analyses will be performed for our secondary outcomes.

Importance: Treatment of obesity-related OSA in adults has been shown to reduce morbidity and mortality. Our study is uniquely poised and timely, as it will be the first to examine the impact of PAP therapy in children on measures of insulin resistance and other obesity-related conditions. It will raise awareness of co-morbidities of obesity and OSA in childhood and support early intervention, before irreversible end-organ damage has occurred.

ELIGIBILITY:
Inclusion Criteria:

* Age 8 to 16 years
* Obesity, defined as body mass index greater than or equal to the 95th percentile for gender and age (2000 CDC Growth Charts for US)
* Moderate to severe OSA diagnosed on polysomnography, for which PAP therapy (continuous positive airway pressure or bi-level positive airway pressure) is prescribed by a physician. Overnight laboratory polysomnography, the gold standard for assessment of OSA115 and titration of PAP, will be performed and scored by a certified sleep technician, according to the American Academy of Sleep Medicine recommendations. Moderate to severe OSA will be defined as an obstructive apneahypopnea index (OAHI) of greater than or equal to 10 apneas or hypopneas per hour. Although no strict guidelines for defining severity of OSA in children exist, the definition for this study was derived by a consensus of pan-Canadian pediatric sleep medicine experts.
* Parents/guardians and children must also be fluent in English or French.

Exclusion Criteria:

* craniofacial anomalies other than tonsillar and adenoid enlargement118, 119
* central nervous system lesions
* neuromuscular, neurological, or genetic syndromes
* congenital heart disease and/or diagnosed ventricular dysfunction
* chronic respiratory disease with the exception of asthma
* use of oral or intravenous corticosteroids within the past 3 months (as this would affect the primary outcome).
* prior exposure to PAP therapy

Ages: 8 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Obese children (body mass index (BMI) ≥ 95th %ile for age and sex) 8-17 years old with moderate-severe OSA will be recruited for this study from four pediatric tertiary care centres across Canada. As per current standard of care, those children with moderate-severe OSA, defined as ≥ 10 obstructive events per hour on polysomnography, will be prescribed PAP treatment.
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-06 (Actual); Primary Completion 2014-07 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
HOMA-IR | 1 year after start of PAP therapy
  Euglycemichyperinsulinemic clamp technique is the gold standard measurement technique for insulin resistance however, invasive and rarely used in clinical practice. A surrogate is the homeostasis model assessment (HOMA) formula for insulin resistance (HOMA-IR) Thus, lower HOMA values indicate higher insulin sensitivity. The estimate obtained with HOMA correlates well with measures of insulin resistance obtained from obese and non-obese children and adolescents with the clamp technique

SECONDARY OUTCOMES:
Systemic Hypertension | 1 year after start of treatment with PAP
  Systemic hypertension,will be measured with 24-hour ABPM at baseline and 1 year. Summary measures for each of the day and night periods include average systolic and diastolic BP, and systolic and diastolic BP loads, as well as % nocturnal dipping. These summary measures have been shown to predict important outcomes including left ventricular hypertrophy, cardiovascular events, and death more accurately than casual BP measures
Heart rate and heart rate variability | 1 year after the start of PAP therapy
  Heart rate and heart rate variability will be analyzed from electrocardiography (EKG) data acquired during polysomnography performed at baseline and 1 year. EKG is more accurate than pulse oximetry to measure high- and low-frequency variability in heart rate and thus is the gold standard for obtaining these measures during sleep.We will focus on the RR interval as a measure of heart rate. Both time-domain components and frequency-domain components will be considered as measures of heart rate variability. We will use normative values as derived by Massin et al.
hsCRP | 1 year after start of PAP therapy
  Blood samples obtained at baseline, 6 months and 1 year will be assessed for levels of CRP, a protein which is released during the chronic inflammation underlying atherosclerosis. Compared with the standard CRP test, the hsCRP assay can detect lower protein concentrations with greater sensitivity and achieves better specificity for predicting vascular events
Conners' Parent and Teacher Rating Scales | 1 Year fter the start fo PAP therapy
  The Conners' Parent and Teacher Rating Scales have demonstrated excellent reliability and validity. These commonly used questionnaires rely on observer ratings to assess attention deficit/hyperactivity disorder (ADHD) and evaluate problem behaviour in children and adolescents. We will use the Revised Short version which contains 27 items with scales measuring oppositional behaviour, cognitive problems/inattention and symptoms of ADHD
Child Behavior Checklist | 1 year after start of PAPA therapy
  The Child Behavior Checklist is one of the most widely-used standardized measures in child psychology for evaluating maladaptive behavioural and emotional problems in children Specifically, this parent-report questionnaire contains 118 items aimed at assessing the frequency of observed internalizing (i.e. anxious, depressive, and overcontrolled) and externalizing (i.e. aggressive,hyperactive, noncompliant, and undercontrolled) behaviors.
Pediatric Quality of Life Inventory (PEDS-QL) | 1 Yaer after start of PAP therapy
  The PEDS-QL is a 23-item test designed to evaluate levels of functioning in 4 areas of health: physical, emotional, social and scholastic. This tool has demonstrated excellent reliability and validity and is frequently used to assess pediatric quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Evelyn Constantin, MD, Principal Investigator — Montreal Children's Hospital of the MUHC; Sherri L Katz, md, Principal Investigator — Childrens Hospital of Eatern Ontario
Locations (4):
- Canada (4):
  - Alberta Children's Hospital, Calgary, Alberta
  - Stollery Children's Hospital, Edmonton, Alberta
  - Childrens Hospital of Eastern Ontario, Ottawa, Ontario
  - Montreal Childrens Hospital, Montreal, Quebec